CLINICAL TRIAL: NCT06485037
Title: Effect of Time-restricted Eating on Appetite and Sleep in Adults With Poor Sleeping Habits
Brief Title: Time-restricted Eating, Appetite and Sleep
Acronym: SLEEPFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TRE-SLEEP-2022
Record Dates: First submitted 2023-10-24; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2023-05

CONDITIONS: Sleep; Appetitive Behavior
Keywords: time-restricted eating; sleep duration; sleep quality; appetite regulation
MeSH Terms: conditions — Appetitive Behavior; Intermittent Fasting; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This was a randomized, controlled experimental study. The recruited participants will be randomized to follow one of two groups: i) TRE, during which the participants will have to restrict the daily time allocated to eating to a window of 10 hours per day but without any other diet modification (e.g., types of food or amount of energy consumed). The fasting period of participants assigned to this intervention must include between 11 p.m. and 6 a.m. Each participant can freely choose the starting time of their eating window. If a participant needs to make modifications to the start time of her feeding window, he/she may do so only once during the study, and the research team must be informed; ii) Control, during which the participants must continue with their usual eating pattern, without making any changes. The duration of the intervention will be 8 weeks. Randomization will be done using computer-generated random numbers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted eating (Experimental): Participants in the TRE group must restrict their eating to a time window of 10 hours per day, with mandatory fasting from 11 p.m. to 6 a.m.
  Interventions: Behavioral: Time-restricted eating
- Control (No Intervention): Participants in the Control group must follow their usual diet routine, without any time restriction

INTERVENTIONS:
Behavioral: Time-restricted eating — Self-selected 10-hour eating window for 2 months
  Arms: Time-restricted eating

SUMMARY:
The goal of this clinical trial is to learn about the effect of time-restricted eating (TRE) to 10 hours per day on the regulation of appetite, the desire to eat, and the quality and duration of nocturnal sleep in adults with normal weight and short sleep duration and/or habitual poor quality sleep.

The main questions it aims to answer are: 1) How does a time-restricted eating protocol affect appetite and desire to eat? and 2) How does a time-restricted eating protocol affect nighttime sleep duration and quality? Participants will be asked to follow a TRE protocol on which they must restrict their eating to a self-selected time window of 10 hours per day (but with mandatory fasting from 11 p.m. to 6 a.m.) for 2 months. Researchers will compare the intervention with a control group, in which the participants should follow their usual diet without any time restriction, to see if the intervention decreases appetite and desire to eat, improves the quality, and increases sleep duration.

DETAILED DESCRIPTION:
Time-restricted eating (TRE) restricts the time to consume food during the day, establishing a feeding window (thus extending the fasting period). It has been suggested that TRE may regulate appetite and sleep quality, even though the evidence is equivocal for these last two aspects. This study aims to determine the effect of TRE (to 10 hours per day) on regulating appetite, the desire to eat, and the quality and duration of nocturnal sleep in normal-weight adults with short-duration and/or habitual poor-quality sleep.

The study sample will be composed of at least 24 participants, randomly assigned to an intervention (TRE) or no-intervention (Control) group. Participants will be recruited in the Santiago Metropolitan region (near the Faculty of Medicine of the University of Chile, Independencia commune) through an open call to participate (through flyers and on social networks). The groups being randomly compared are: i) TRE (intervention group), in which participants must restrict their eating to a time window of 10 hours per day, with mandatory fasting from 11 p.m. to 6 a.m.; and ii) Control (no-intervention group), in which the participants should follow their usual diet, without any time restriction. Both groups will be evaluated before, during, and after 2 months.

In both groups, the following main parameters will be evaluated: i) appetite and satiety feelings (through visual analog scales) and the intense desire to eat (through a Food Craving inventory); ii) the quality of habitual sleep during the last month (through the Pittsburgh Sleep Quality Index) and, nighttime sleep duration (through 7-days actigraphy recordings); iii) diet composition and quality (through 24-h recall). Measurements of anthropometry and body fat will also be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Young (age between 18 to 45 years)
* Healthy adults
* Both women and men
* Body-mass index between 18.5 to 24.9 kg/m2
* Report sleeping less than 7 hours per night and/or who have poor sleep quality.

Exclusion Criteria:

* Night shift workers
* Patients with psychiatric disorders
* Patients with neurological diseases
* Patients with uncontrolled thyroid disease
* Lactating and pregnant women
* Patients with type-1 or type-2 diabetes
* Persons with high blood pressure or hypertension
* Patients with uncontrolled dyslipidemia
* Patients with sleep disorders
* Persons who perform intense physical exercise more than 3 times a week

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Appetite feeling as assessed by a Visual Analog Scale | 2 months
  A visual analog scale was used to assess appetite feeling. Each participant rates their subjective feelings of appetite (before and after completion of the study) using a 100 mm visual analog scale, with endpoints indicating from "not at all" (0 mm) to "extremely" (100 mm).
Satiety feeling as assessed by a Visual Analog Scale | 2 months
  A visual analog scale was used to assess satiety feeling. Each participant rates their subjective feelings of satiety (before and after completion of the study) using a 100 mm visual analog scale, with endpoints indicating from "not at all" (0 mm) to "extremely" (100 mm).
Sleep quality as assessed by the Pittsburgh Sleep Quality Index | 2 months
  The Pittsburgh Sleep Quality Index (PSQI) was used to assess sleep quality. The PSQI is a 19-item questionnaire evaluating subjective sleep quality over the previous month. Each participant rated each of the 19 questions (before and after completion of the study), and the questions were combined into 7 clinically-derived component scores. The 7 component scores are added to obtain a global score ranging from 0-21, with higher scores indicating worse sleep quality. Sleep quality score was also categorized as good sleep quality (a global score of less than 5 points) and poor sleep quality (a global score ≥ 5 points).
Sleep duration as assessed by actigraphy | 2 months
  The actigraphy technique measured habitual sleep duration and sleep pattern. Each participant used the Actiwatch®64 (Respironics Mini Mitter Company, Inc.) actigraph for 7 consecutive days on the non-right-handed wrist (before and after completion of the study). The mean total sleep duration (in minutes) is obtained for the recording days.

SECONDARY OUTCOMES:
Craving for foods as assessed by the Food Craving inventory | 2 months
  The Food craving inventory assessed the intense desire (craving) to eat a food. Each participant rated their subjective craving for specific foods, scored from 0 to 4 (where 0 = never; 1 = rarely; 2 = sometimes; 3 = often; and 4 = always/almost every day) according to the strength of the craving. Foods are grouped into four groups: high-fat foods, sweets, carbohydrates/starches, and fast-food fats. A global craving score and four food-specific subscores were obtained.
Energy intake as assessed by 24-hour dietary recall | 2 months
  A 24-hour dietary recall (24hDR) was used to assess each participant's dietary intake (before and after completion of the study). The 24hDR was applied to each participant. Diet composition was obtained from the USDA National Nutrient Database for Standard Reference and a local (Chilean) database. The total daily energy (expressed as kcal/day) and macronutrient (protein, carbohydrate, and fat; expressed as g/day) intake was obtained through the software Food Processor SQL® (ESHA Research, Salem, OR, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Chamorro, Dr, Principal Investigator — Department of Nutrition, University of Chile
Locations (1):
- Department of Nutrition, University of Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
Published data generated from the study will be available from the leading author, upon reasonable request.

REFERENCES:
- [Derived] Beaumont A, Farias R, Fernandez W, Lizama C, Gonzalez J, Villar A, Varady KA, Peirano P, Chamorro R. Time-restricted eating improves appetite regulation and sleep characteristics in adults with poor sleep quality. Clin Nutr. 2025 Jul;50:66-74. doi: 10.1016/j.clnu.2025.04.028. Epub 2025 May 2. PMID 40373727